CLINICAL TRIAL: NCT05364216
Title: Effect of Thoracic Paravertebral Block on Chronic Pain and Cognitive Function After Thoracoscopic Partial Pulmonary Resection in Elderly Patients
Brief Title: Effect of TPVB on Postoperative Pain and Cognitive Function After VATS in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20220503
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Cognitive Dysfunction; Acute Postoperative Pain; Chronic Postsurgical Pain
Keywords: Thoracic paravertebral block; Cognitive function; Chronic Postsurgical Pain
MeSH Terms: conditions — Postoperative Cognitive Complications; Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Other): The general anesthesia was used.In this group, cognitive function was evaluated by MMSE and MoCA scale on one day before surgery, one day after surgery, and three months after surgery. Acute postoperative pain was was evaluated by VAS after extubation , one day after surgery, Chronic postsurgical pain was evaluated by VAS on three months after surgery.
  Interventions: Behavioral: Measurement of cognitive function
- Group T (Experimental): Group T received 0.375% ropivacaine 20ml thoracic paravertebral nerve block combined with general anesthesia under ultrasound guidance after anesthesia induction.
  Interventions: Behavioral: Measurement of cognitive function; Procedure: Thoracic paravertebral block
- Non-surgical controls (Other): Age and sex-matched community people are included for three sessions of MMSE test evaluation for calculation of POD incidence as normal control to in Z value calculation of POD incidence to rule out learning effect.
  Interventions: Behavioral: The assessment of cognitive function

INTERVENTIONS:
Behavioral: Measurement of cognitive function — Patients undergoing thoracoscopic surgery underwent general anesthesia.MMSE and MoCA were assessed at one day before surgery, one day after surgery, and three months after surgery
  Other Names: assessment of POD
  Arms: Group C; Group T
Procedure: Thoracic paravertebral block — The patient was placed in lateral supine position, and the T5 spinous process was moved 2 to 3 cm laterally to the operative side as the puncture point, and the pleura and T5 transverse process were observed, and the paraspinal space was observed on the lower lateral side of the transverse process. Using in-plane technique, the needle position was adjusted under ultrasound visualization to reach the paraspinal space. 20ml 0.375% ropivacaine was injected into the suction syringe when there was no blood or gas, and the drug liquid could be seen spreading outside the pleura. "Landscape sign" appeared, indicating successful block
  Other Names: General anesthesia
  Arms: Group T
Behavioral: The assessment of cognitive function — Participants were assessed for MMSE and MoCA at the same period as the group C
  Arms: Non-surgical controls

SUMMARY:
To investigate the effect of ultrasound-guided thoracic paravertebral nerve block on postoperative acute and chronic pain and cognitive function in elderly patients with thoracoscopic partial lung resection.

DETAILED DESCRIPTION:
A total of 92 patients who were admitted to Qinhuangdao First Hospital for and divided into control group (group C ), thoracic paravertebral nerve block combined with general anesthesia group (group T).

Group C received general anesthesia, and group T received 0.375% ropivacaine 20 ml of thoracic paravertebral nerve block combined with general anesthesia after induction of anesthesia. SBP（Systolic Blood Pressure）/DBP （Diastolic Pressure）and HR（Heart Rate） of the two groups were recorded before anesthesia induction (T1), at the time of intubation (T2), at the beginning of surgery (T5), immediately after surgery (T6), and five minutes after extubation (T7) . rScO2（Regional cerebral oxygen saturation） was recorded in both groups at (T1), five minutes after induction(T3), five minutes after single lung ventilation on lateral recumbent(T4), (T6), (T7). The incidence of acute and chronic pain after surgery was compared between the two groups by NRS（Numerical Rating Scale）after extubation , one day after surgery, and three months after surgery.

The cognitive function of the two groups was assessed with the Mini Mental State Scale (MMSE) and the Montreal Cognitive Assessment Scale (MoCA-Beijing) on the day before , one day after and three months after surgery, comparing the incidence of PND (postoperative cognitive dysfunction) between the two groups.Analyze whether paravertebral block can reduce the incidence of POD by improving brain oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 30 kg/m2
* American Society of Anesthesiologists (ASA) grades I-III
* The score of Mini Mental state examination≥24
* The score of Montreal Cognitive Assessment-Beijing Scale≥26

Exclusion Criteria:

* Patients with heart, lung, brain and other vital organ disorders
* The score of Mini Mental state examination≤23
* The score of Montreal Cognitive Assessment-Beijing Scale≤25
* Preoperative psychiatric disorders or long-term use of drugs affecting the psychiatric system
* Have severe visual, hearing, speech impairment or other inability to communicate with the visitor
* Have contraindications to thoracic parathymic block
* Refuse to sign informed consent

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of POD at one day after surgery | One day after surgery
  The MMSE and MoCA difference between the patients on the day before surgery and one day after surgery was compared and substituted into the formula.The formula of Z-scoring method is Z= (XC-X) /SDXC, where X refers to the change value of patients' MMSE/MoCA score at one day before surgery and one day after surgery. XC is the mean change value of the non-surgical control group at the same time, and SDXC is the standard deviation of the change value of the non-surgical control group. Finally, the Z-value at one day after surgery is calculated respectively. If the value of Z is ≥1.96, the patient is considered to have developed POCD
Incidence of POD at three months after surgery | Three months after surgery
  The MMSE and MoCA difference between the patients on the day before surgery and three months after surgery was compared and substituted into the formula.The formula of Z-scoring method is Z= (XC-X) /SDXC, where X refers to the change value of patients' MMSE score at one day before surgery and three months after surgery. XC is the mean change value of the non-surgical control group at the same time, and SDXC is the standard deviation of the change value of the non-surgical control group. Finally, the Z-value at three months after surgery is calculated respectively. If the value of Z is ≥1.96, the patient is considered to have developed POCD
Change in pain assessed by Visual Analogue Scale | Five minutes after extubation
  Divide the ruler into 10 equal parts, with 0 means no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain(Patients have mild restrictions on daily activities or mild sleep disturbances due to pain，maybe require additional analgesic treatment), and 7-10 indicating severe pain(Patients are unable to fall asleep and cannot perform daily activities，they strongly request the use of analgesics).
Change in pain assessed by Visual Analogue Scale | One day after surgery
  Divide the ruler into 10 equal parts, with 0 means no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain(Patients have mild restrictions on daily activities or mild sleep disturbances due to pain，maybe require additional analgesic treatment), and 7-10 indicating severe pain(Patients are unable to fall asleep and cannot perform daily activities，they strongly request the use of analgesics).
Change in pain assessed by Visual Analogue Scale | Three months after surgery
  Divide the ruler into 10 equal parts, with 0 means no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain(Patients have mild restrictions on daily activities or mild sleep disturbances due to pain，maybe require additional analgesic treatment), and 7-10 indicating severe pain(Patients are unable to fall asleep and cannot perform daily activities，they strongly request the use of analgesics).

SECONDARY OUTCOMES:
The change of SBP/DP | before anesthesia induction , at the time of intubation , at the beginning of surgery , immediately after surgery , and five minutes after extubation
  The change of Systolic blood pressure(SBP) and Diastolic pressure(DP) among the two groups
The change of HR | before anesthesia induction , at the time of intubation , at the beginning of surgery , immediately after surgery , and five minutes after extubation
  The change of Heart rate(HR) among the two groups
The change of rScO2, maximum and minimum of rScO2, duration of 10% below the base value | before anesthesia induction , five minutes after induction, five minutes after single lung ventilation on lateral recumbent, immediately after surgery, and five minutes after extubation
  The change of regional cerebral oxygen saturation(rScO2), maximum and minimum of rScO2, duration of 10% below the base value among the two groups
Anesthetic drug | during the surgery
  The dosage of remifentanil and propofol in different groups were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Qinshuang Liu, master, Study Director — The First hosptial of Qinhuangdao; Linyu Shi, master, Study Chair — The First hosptial of Qinhuangdao
Locations (1):
- The First hosptial of Qinhuangdao, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: No